CLINICAL TRIAL: NCT02922517
Title: Predictive Factors and Consequences of Myocardial Fibrosis in Hypertrophic Cardiomyopathy
Acronym: HCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Lille (Other); Rennes University Hospital (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: Prog/11/35
Record Dates: First submitted 2013-03-25; First posted 2016-10-04 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: biomarkers; echocardiography; MRI imaging; nuclear medicine
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for biomarkers assessment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with obstructive HCM: patients with HCM (obstructive or no obstructive)
- controls: patients without HCM
- patients with non obstructive HCM: patients with non obstructive HCM

SUMMARY:
Fibrosis, myocardial deformation and biomarkers in hypertrophic cardiomyopathy (HCM)

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a rare genetic disease (1), whose phenotypic expression is found in less than 1/1000 people, mainly linked to a mutation of a protein of the sarcomere (14 genes and 400 mutations identified nowadays). HCM occurs in about 50% of cases in young adults under the age of 30 years. Progress in the identification of the responsible mutation does not have allowed significant advances for the clinical management and evaluation of the prognosis of patients with HCM. In fact, the link between genotype and phenotype is poor in the HCM, so that identification of the mutation in approximately 60% of patients does not properly characterize the disease and its evolution. It is therefore necessary to identify new markers to better characterize HCM patients. Myocardial fibrosis could be a severity marker of the HCM but its consequences and determinants are little known or unknown.

The objective of this work is to identify the determinants and consequences of myocardial fibrosis in HCM, particularly the relationship between fibrosis and left ventricular dysfunction assessed by the analysis of myocardial deformation and between fibrosis and heart failure. The study of fibrosis, which concerns 30 to 70% of patients and replace 1 to 70% of the myocardial tissue, is made possible in vivo by analysis of delayed enhancement gadolinium in MRI. This work aims to study the relationship between myocardial fibrosis, heart function assessed by myocardial deformation, heart failure, and biological profile (proteomics) of patients at rest and after exertion.

This study is an observational research. Indeed, all examinations are done as part of usual care patients. Only additional tubes of blood are collected in the initial biological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known HCM or recently discovered with a wall thickness greater than or equal to15 mm without family background or> 13 mm in an HCM family context in the absence of other causes found capable of producing such a degree of hypertrophy
* HCM apparently linked to a mutation of a protein of the sarcomere (identified mutation or absence of other causes of hypertrophy found when the mutation search was not performed or was unsuccessful)
* Control subjects will be patients greater than or equal to 18 years without known cardiovascular disease or that may affect their ability to function, addressed to achieve a stress echocardiography for assessment of atypical symptoms, with a low pretest probability of coronary artery disease, and accepting blood sample before and after exercise. They do not realize Holter ECG or cardiac MRI as part of the study.

Exclusion Criteria:

* Refusal of the patient
* Age < 16 years old
* Valvulopathy associated significant (grade 3 or 4 regurgitation, or severe stenosis) other than mitral insufficiency
* Defibrillator, pacemaker, or other cons-indication or intolerance to achieving MRI
* Unable to receive clear information (patient's intellectual default)
* Under protective measure of justice

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sex over 16 year-old with HCM
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
measurement of the overall longitudinal myocardial strain (in 2D strain) | day 90

SECONDARY OUTCOMES:
global myocardial longitudinal deformation (three-dimensional) | day 90
Transforming growth factor (TGF) blood dosage | at year 3
Bone morphogenetic protein 2 (BMP2) blood dosage | at year 3
Periostin blood dosage | at year 3
Heart Failure Symptoms evaluation | day 90
  New York Heart Association (NYHA) stage, presence of congestive signs according to the Framingham Heart Study, functional capacity
type of heart failure | day 90
  sub aortic obstruction if gradient rest or effort greater than or equal to 30 mmHg, left ventricle (LV) systolic dysfunction assessed on the ejection fraction (EF) less than or equal to 50%, restrictive heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mabo, PU-PH, Principal Investigator — Rennes University Hospital; Erwan Donal, McU-PH, Principal Investigator — Rennes University Hospital; Pascal de Groote, PH, Principal Investigator — Lille University Hospital; Anne-Sophie Polge, PH, Principal Investigator — Lille University Hospital; Marjorie Richardson, PH, Principal Investigator — Lille University Hospital; Nicolas Lamblin, PH, Principal Investigator — Lille University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France